CLINICAL TRIAL: NCT05269927
Title: A Multi-domain Approach for the Characterization and Early Diagnosis of Neurodevelopmental Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Eugenio Medea (Other)
Collaborators: Ministry of Health, Italy (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 707
Record Dates: First submitted 2022-02-01; First posted 2022-03-08 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Neurodevelopmental Disorders
Keywords: Neurodevelopmental disorder; EEG; Multi-domain data; Machine Learning
MeSH Terms: conditions — Neurodevelopmental Disorders | interventions — Electroencephalography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TD (typically developing) infants (Experimental): Typically developing infants, infants without familiar risk for ASD or LD.
  Interventions: Diagnostic Test: EEG; Diagnostic Test: DNA samples; Diagnostic Test: clinical data; Other: environmental data
- HR (high risk) for LD infants (Experimental): Infants at high risk for language disorders
  Interventions: Diagnostic Test: EEG; Diagnostic Test: DNA samples; Diagnostic Test: clinical data; Other: environmental data
- HR for ASD infants (Experimental): Infants at high risk for autism spectrum disorder
  Interventions: Diagnostic Test: EEG; Diagnostic Test: DNA samples; Diagnostic Test: clinical data; Other: environmental data

INTERVENTIONS:
Diagnostic Test: EEG — resting state EEG
Diagnostic Test: DNA samples — genotypings of twelve CNTNAP2 SNPs from DNA obtained by saliva samples
Diagnostic Test: clinical data — standardized scales measuring the infants' cognitive, motor and linguistic development administered at 6, 12 and 18. Measures available at 6 and 12 months: a) Bayley Scales of Infant and Toddler Development- Third Edition; b) Griffiths mental development scales (0-2) (GMDS-R); Measures available at 18 months: c) Language Development Survey (LDS); d) "Il PRIMO VOCABOLARIO DEL BAMBINO" (PVB); e) CHILD BEHAVIOR CHECKLIST (CBCL); (f) Modified Checklist for Autism in Toddlers (M-CHAT).
Other: environmental data — questionnaires administered to parents related to the following environmental factors: a) information about the presence of a clinical diagnosis of neurodevelopmental disorders within first-degree relatives; b) gestational age; c) birth weight; d) parental age and education; e) socio-economic status

SUMMARY:
Diagnosis and characterization of neurodevelopmental disorders are considered challenging processes because of their complexity, multi-factoriality and heterogeneity. The present project will consider two of the most common neurodevelopmental disorders (i.e. autism spectrum disorders (ASD) and language disorders (LD)), with the aim to overcome these difficulties, by: a) deeply investigating their neuronal correlates; b) identifying multi-domain biomarkers (electrophysiological, genetic, environmental and clinical); c) developing a machine learning algorithm for early diagnosis. To achieve the above mentioned aims a multi-domain dataset will be used, comprising data collected from typically developing infants, infants at high risk for ASD and infants at high risk for LD. The data that will be used have been already collected within other trials performed at the Scientific Institute E. Medea.

ELIGIBILITY:
Inclusion Criteria:

* APGAR scores at birth at 1' and 5' > 7;
* newborn screening otoacoustic emissions in the norm;
* absence of neurological disorders;
* Italian as the language mainly spoken in the family nucleus.

Exclusion Criteria:

* APGAR scores at birth at 1' and 5' <= 7;
* newborn screening otoacoustic emissions not in the norm;
* presence of neurological disorders;
* non-Italian native speaker

Ages: 5 Months to 7 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
EEG power spectral density (PSD) | one year after the end of the recruitment
  Power spectral density (PSD) estimated in the delta, theta, alpha, beta and gamma frequency bands of the EEG
EEG signal coherence | 18 months after the end of the recruitment
  EEG signal coherence
EEG signal entropy | 18 months after the end of the recruitment
  EEG signal entropy

CONTACTS AND LOCATIONS:
Locations (1):
- Scientific Institute IRCCS E. Medea, Bosisio Parini, Lecco, Italy